CLINICAL TRIAL: NCT04908995
Title: A Single-Center, Double-Blind, Placebo-Controlled, Phase 1a, Fed-Fasted, Crossover Study To Investigate The Safety, Tolerability, Pharmacokinetics, And Food Effects Of A Single Oral Dose Of EC5026 In Healthy Male And Female Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Food Effects of Oral EC5026 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EicOsis Human Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC5026-1-03
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy Adults
MeSH Terms: interventions — EC5026

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EC5026 (Experimental): Single 8 mg oral dose of EC5026
  Interventions: Drug: EC5026 oral tablet
- Placebo (Placebo Comparator): Single dose of matching oral placebo
  Interventions: Other: Placebo oral tablet

INTERVENTIONS:
Drug: EC5026 oral tablet — 12 subjects will receive a single oral 8 mg dose of EC5026 in two Dosing Periods (one in fed state and one in fasted state) separated by a Washout Period. Subjects in this group will be randomized 1:1 to one of 2 sequences:
  * Dosing Sequence A: Subjects will be dosed in a fed state in Dosing Period 1 and in a fasted state in Dosing Period 2, or
  * Dosing Sequence B: subjects will be dosed in a fasted state in Dosing Period 1 and in a fed state in Dosing Period 2.
  Arms: EC5026
Other: Placebo oral tablet — 6 subjects will receive an oral dose of matching placebo in one single Dosing Period. Subjects in this group will be randomized 1:1 to receive placebo under fed or fasted conditions.
  Note: Subjects assigned to the placebo arm will not return for a second Dosing Period.
  Arms: Placebo

SUMMARY:
The purpose of the study is to provide safety, tolerability, pharmacokinetics and food effects data of a single 8 mg oral dose of EC5026 in healthy subjects.

DETAILED DESCRIPTION:
This is a single-center, double-blind, placebo-controlled, Phase 1a single dose study fed-fasted study evaluating the safety, tolerability, pharmacokinetics and food effects of a single 8 mg oral dose of EC5026 in healthy male and female subjects. EC5026 is an inhibitor of the soluble Epoxide Hydrolase (sEH) enzyme developed as a first-in-class analgesic for the treatment of pain. This study will help refine the dosing strategy for subsequent multiple-dose studies in healthy subjects and for future clinical trials in patients with pain.

sEH is an enzyme that is downstream in the cytochrome P450 (CYP) pathway of the arachidonic acid (AA) cascade. The sEH enzyme is responsible of metabolizing a class of epoxy-fatty acids known as epoxyeicosatrienoic acids (EETs), which are potent, naturally occurring analgesics. EETs are produced at high concentrations in areas of tissue damage and inflammation, but are rapidly metabolized by the sEH enzyme into inactive compounds. Effective inhibition of sEH activity prolongs the ability of EETs to exert their analgesic activity.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Males or females must be 18-70 years of age.
2. Subjects must be willing to provide written informed consent to participate in the study.
3. Subjects must be in generally good health as determined by prestudy medical history, physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG).
4. Subjects must be willing to remain in confinement at the CRU for up to 4 consecutive days in 2 separate dosing periods and to return to the unit as specified for additional blood tests and safety evaluations during the study period.
5. Subjects must have a body mass index of 19-32 kg/m2.
6. Subjects must have a normal blood pressure (systolic blood pressure 90-140 mm Hg, diastolic blood pressure 50-90 mm Hg) and heart rate (resting heart rate 45-90 beats per minute) without medication. Blood pressure and heart rate may be repeated at the discretion of the investigator. If the value continues to be out of range but not clinically significant, the subject may continue per the discretion of the investigator.
7. Subjects must have a clinical chemistry profile, including electrolytes, alkaline phosphatase (ALP), lactate dehydrogenase, creatine phosphokinase (CPK), creatinine, and urea, within the normal range without medication at screening. Subjects who have mildly out of range laboratory results that are not considered clinically significant by the investigator can be included in the study.
8. Subjects must have an early morning (collected between 0600 AM and 0800 AM) serum cortisol level >10 mcg/dL (>275.9 nmol/L) and early morning adrenocorticotropic hormone (ACTH) and aldosterone levels within the normal range at screening.
9. Subjects must be nonsmokers or willing to abstain from smoking 2 weeks prior to randomization and for the duration of the study.
10. Subjects must be able to read, understand, and follow the study instructions.
11. Male subjects and their female sexual partners must agree to use double-barrier contraception during the study period and for 2 months after clinic discharge or to provide proof of postmenopausal state (minimum 1 year) or surgical sterility. Surgical sterility will be defined as proof of female sterilization (via tubal ligation, bilateral salpingo-oophorectomy or hysterectomy) or male sterilization (vasectomy, with laboratory proof of postvasectomy sterilization assessed at least 16 weeks postprocedure).
12. Male subjects must not donate sperm during the study and for 12 months after receiving the last dose of study drug.
13. Female subjects must be nonpregnant, nonlactating, and either postmenopausal for at least 1 year, or surgically sterile for at least 3 months, or they must agree to use double barrier contraception from 28 days and/or their last confirmed menstrual period prior to study enrollment (whichever is longer) until 2 months after clinic discharge. Double-barrier contraception may include, but is not limited to, nonhormonal intrauterine device with spermicide, female condom with spermicide, diaphragm with spermicide, cervical cap with spermicide; having a male sexual partner who agrees to use a male condom with spermicide; or having a sterile sexual partner. Females on hormonal contraceptives ( including hormonal intrauterine device or oral contraceptives) will be excluded from the study. For all females of childbearing potential, the pregnancy test result must be negative at screening and prestudy baseline (Day -1).

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subjects with any abnormalities in any of the following: liver function tests, CPK, or urinalysis results. Liver function tests, CPK, or urinalysis tests may be repeated at the discretion of the investigator, if necessary, to confirm any abnormalities. Subjects who have mildly out of range CPK or urinalysis results that are not considered clinically significant by the investigator can be included in the study.
2. Subjects who have used any nonstudy medication(s), including low-dose aspirin for cardiovascular prophylaxis, within 1 week before administration of study drug. This includes any drug that can confound the results of the food-effect study, such as drugs that can alter the absorption of other drugs by affecting gastrointestinal motility or by changing the gastric pH, as well as drugs that can increase or decrease the metabolism and excretion of other drugs.
3. Subjects who have used chemotherapy agents or who have a history of cancer, other than nonmetastatic skin cancer that has been completely excised, within 5 years prior to screening.
4. Subjects with a history of bacterial, fungal, or viral infection requiring treatment with antibiotics, antifungal agents, or antivirals within 1 month prior to randomization.
5. Subjects with a history of disorders of the hypothalamic-pituitary-adrenal (HPA) or hypothalamic-pituitary-gonadal (HPG) axis.
6. Subjects with a presence or history of peripheral edema within the past 5 years.
7. Subjects with a history of congestive heart failure.
8. Subjects who have used (within 30 days of randomization) or plan on using any of the following during the duration of the study

   1. any prescription or over-the-counter drugs that are cytochrome P450 (CYP) inducers or inhibitors (e.g., cimetidine, paroxetine, fluoxetine, haloperidol, ketoconazole, itraconazole, fluconazole, erythromycin, or clarithromycin)
   2. any dietary aids, supplements, or foods that are known to modulate drug metabolizing enzymes (eg, St. John's wort, grapefruit juice).
9. Subjects who have used long term, high-dose, systemic glucocorticosteroids in the previous year or long term topical glucocorticosteroids.
10. Subjects with difficulty in swallowing oral medications.
11. Subjects with a history of seizure disorder (excluding childhood febrile seizure).
12. Subjects with serious psychosocial comorbidities as determined by the principal investigator.
13. Subjects with current cognitive or major psychiatric disorders or any other condition that could interfere with compliance with study procedures and/or confinement in a CRU.
14. Subjects with a positive drug or alcohol test during screening and/or admission.
15. Subjects who have used any other investigational drug within 1 month prior to first study drug administration.
16. Subjects who have used prescription drugs within 1 month or 5 half-lives, whichever is longer, prior to randomization.
17. Subjects who have used any over-the-counter medications, excluding routine vitamins, but including megadose vitamin therapy, within 1 week of enrollment.
18. Subjects who have donated and/or received any blood or blood products (more than 450 mL) within 3 months prior to enrollment.
19. Subjects with a presence or history of active gastrointestinal, renal, hepatic, or coagulant disorder within 1 month prior to enrollment.
20. Subjects with a presence or history of esophageal or gastroduodenal ulceration within 1 month prior to enrollment.
21. Subjects with a family history of significant cardiac disease (ie, sudden death in first degree relative; myocardial infarction prior to 50 years old).
22. Subjects with confirmed coronavirus disease 2019 (COVID-19) (test positive for severe acute respiratory syndrome coronavirus 2 [SARS CoV-2]) or suspected COVID-19 (eg, developed symptoms of a respiratory infection, such as cough, sore throat, shortness of breath, or fever but did not get tested for COVID-19) or known history of COVID-19 within 6 months prior to study entry.
23. Subjects who receive immunization for SARS-CoV-2 within 30 days of randomization or are planning to receive it during the duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAE) [Safety and Tolerability] | 77 days
  All AEs reported or observed during the study will be recorded on the electronic case report forms (eCRF). Information to be collected includes drug treatment, type of event, time of onset, dosage, investigator-specified assessment of severity and relationship to study drug, time of resolution of the event, seriousness, any required treatment or evaluations, and outcome. Any AEs resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. All AEs will be followed until they are resolved, stable, or judged by the investigator to be not clinically significant. The Medical Dictionary for Regulatory Activities will be used to code all AEs.
Area under the plasma concentration versus time curve (AUC) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Maximum observed plasma concentration (Cmax) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Time to maximum observed plasma concentration (Tmax) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Terminal elimination rate constant in plasma (Kel) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Terminal phase half-life in plasma (t1/2) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Apparent total body clearance (CL/F) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Apparent volume of distribution based on the terminal elimination rate constant in plasma (Vz/F) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Renal clearance (CLR) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Amount of drug excreted unchanged in urine (Ae) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Amount of drug excreted within the time interval t1 to t2 (Ae(t1-t2)) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.
Fraction of eliminated dose in urine (Fe%) in response to a single 8mg EC5026 oral tablet [Plasma Pharmacokinetics]. | 14 days
  Standard noncompartmental methods will be used. The effects on this parameter of a effect of a high-fat, high-calorie meal will be evaluated in comparison to fasted conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No